CLINICAL TRIAL: NCT01094158
Title: A Phase II Placebo Controlled Randomised Study of Aramchol on Liver Triglyceride in Patients With Steatosis Due to NAFLD or NASH
Brief Title: Study of Aramchol in Patients With Fatty Liver Disease or Nonalcoholic Steatohepatitis
Acronym: Aramchol003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galmed Medical Reserch (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Beilinson Hospital, Petach Tikva,Israel (Unknown); Meir Medical Center (Other); Kaplan Hospital ,Rehovot,Israel (Unknown); Soroka Hospital,Beer Sheva,Israel (Unknown); Hadassah Medical Organization (Other); Hillel Yaffe Medical Center (Other Government); Rambam Hospital, Haifa, Israel (Unknown); The Lady Davis Carmel Medical Center (Unknown); Holy Family Hospital, Nazareth, Israel (Other); Ziv Hospital (Other Government)
Responsible Party: Doctor Ran Oren, Liver unit, Department of Gastroenterology and Hepatology, Sourasky Medical Center. Tel Aviv.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Aramchol NAFLD Phase-II
Record Dates: First submitted 2010-02-17; First posted 2010-03-26 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Metabolic Syndrome
Keywords: NAFLD; NASH; Fatty Liver; Metabolic Syndrome; Endothelial Dysfunction; Insulin Resistance; Liver Fat
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Fatty Liver; Insulin Resistance | interventions — aramchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high dose (Experimental): Aramchol 300 mg daily (high dose)
  Interventions: Drug: Aramchol
- low dose (Experimental): 100 mg daily (low dose)
  Interventions: Drug: Aramchol
- Placebo (Placebo Comparator): Placebo and two doses will be compared. The Aramchol: placebo ratio is of 2:1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aramchol — 100mg/d tablets packaged in bottles given orally once a day in the morning within 10 minutes after breakfast for a total period time of 3 months
  Other Names: Arachidyl amido cholanoic acid
  Arms: low dose
Drug: Aramchol — 300 mg/d tablets packaged in bottles given orally once a day in the morning within 10 minutes after breakfast for a total period time of 3 months
  Other Names: Arachidyl amido cholanoic acid
  Arms: high dose
Drug: Placebo — tablets packaged in bottles given orally once a day in the morning within approximately 10 minutes after breakfast
  Arms: Placebo

SUMMARY:
Primary purpose: Compare the changes in liver triglycerides concentration in the Aramchol versus the placebo arm following three month treatment.

Secondary purpose: Comparing liver enzymes, markers of endothelial dysfunction, insulin resistance, SCD1 activity and cholesterol synthesis and lipid levels, between the Aramchol and the placebo arms.

DETAILED DESCRIPTION:
A Phase II, multicenter, double blind, randomized, placebo controlled study on the effect of Aramchol on liver triglycerides concentration in patients with steatosis due to NAFLD or NASH

The purpose of the study is to test whether Aramchol will reduce safely and effectively liver fat concentration in patients with NAFLD and NASH.

Aramchol inhibits the liver enzyme Stearoyl Coenzyme A Desaturase (SCD). It reduces fatty acid synthesis while increasing fatty acid oxidation. It was shown to reduce liver fat in animal models with diet induced Fatty Liver. It has also marked hypocholesterolemic effects, mainly via upregulation of theABCA1 cholesterol transporter. It thus causes(incomplete) SCD inhibition while being antiatherogenic

Primary purpose: Compare the changes in liver triglycerides concentration in the Aramchol versus the placebo arm following three month treatment.

Secondary purpose: Comparing liver enzymes, markers of endothelial dysfunction, insulin resistance, SCD1 activity and cholesterol synthesis and lipid levels, between the Aramchol and the placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven NAFLD or NASH based on a biopsy performed during the preceding 18 months fulfilling the following criteria:

  * At least 15% of hepatocytes showing steatosis,with Fibrosis of not more than stage 3, with at most bridging fibrosis.

Patients with a NAFLD activity score 0-2 will be considered to have NAFLD. Biopsies with an activity score of 3 or more will be considered NASH.

* Triglycerides concentration in the liver of 6% or more as measured by NMRS.
* At least two elevated serum ALT levels in the previous six months, with latest test within 2 months of trial.
* Normal or only slightly impaired synthetic liver function (serum albumin >3.5gm%, INR 0.8-1.3)
* Male or female aged 18-75 years.
* Negative pregnancy test at study entry for females of child bearing potential.
* Females of child bearing potential practicing reliable contraception throughout the study period.
* Signature of the written informed consent

Exclusion Criteria:

* Evidence of cirrhosis on liver biopsy.
* Evidence of fibrosis of more than stage 3 on liver biopsy.
* Patient with liver disease due to acute or chronic hepatitis A, B,C, HIV, and all other liver diseases affecting liver function. Patients with cysts, hemangiomas, or similar abnormalities, are accepted.
* BMI > 35 or >130 kg body weight
* Any other concomitant, significant: metabolic, infectious, inflammatory, neoplastic, or other non-liver disease.
* Various concomitant diseases requiring chronic steroid administration.
* Use of warfarin, metformin, thiaglitazones, insulin or current steroid therapy of more than 3 days.
* Use of other investigational agents < 30 days prior to the study.
* Pregnancy
* Daily alcohol intake > 10gm/day.
* Patients with symptoms of significant mental illness. Inability to cooperate or communicate with the investigator, who are unlikely to comply with the study requirements, or who are unable to give informed consent.
* Performance status: WHO performance status ≥4.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The difference between initial and final liver triglyceride concentration (measured by NMRS) comparing the Aramchol and placebo treated patients. | 3 months

SECONDARY OUTCOMES:
Comparing secondary variables of liver, metabolic and endothelial functions between the Aramchol and the placebo arms. | 3 months
  Comparing liver enzymes, markers of endothelial dysfunction, insulin resistance, SCD1 activity and cholesterol synthesis and lipid levels, between the Aramchol and the placebo arms

CONTACTS AND LOCATIONS:
Overall Officials: Ran Oren, Doctor, Principal Investigator — Liver & Gastroenterology Department,The Tel Aviv Sourasky Medical Center
Locations (11):
- Israel (11):
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah Ein Kerem M.C, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Holy Family HOSPITAL, Nazareth
  - Belinson,Rabin Medical Center, Petah Tikva
  - Kaplan M.C, Rehovot
  - Safed Ziv Hospital, Safed
  - The Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Background] Leikin-Frenkel A, Goldiner I, Leikin-Gobbi D, Rosenberg R, Bonen H, Litvak A, Bernheim J, Konikoff FM, Gilat T. Treatment of preestablished diet-induced fatty liver by oral fatty acid-bile acid conjugates in rodents. Eur J Gastroenterol Hepatol. 2008 Dec;20(12):1205-13. doi: 10.1097/MEG.0b013e3282fc9743. PMID 18989145
- [Background] Gilat T, Leikin-Frenkel A, Goldiner I, Juhel C, Lafont H, Gobbi D, Konikoff FM. Prevention of diet-induced fatty liver in experimental animals by the oral administration of a fatty acid bile acid conjugate (FABAC). Hepatology. 2003 Aug;38(2):436-42. doi: 10.1053/jhep.2003.50348. PMID 12883488
- [Derived] Safadi R, Konikoff FM, Mahamid M, Zelber-Sagi S, Halpern M, Gilat T, Oren R; FLORA Group. The fatty acid-bile acid conjugate Aramchol reduces liver fat content in patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2014 Dec;12(12):2085-91.e1. doi: 10.1016/j.cgh.2014.04.038. Epub 2014 May 9. PMID 24815326